CLINICAL TRIAL: NCT01250691
Title: Epidemiologic Study of Hospital Acquired Pneumonia in a Respiratory ICU
Brief Title: Effects of Isolated Rooms on the Prevalence of Hospital Acquired Pneumonia in a Respiratory ICU
Status: Completed | Type: Observational
Sponsor: Eskisehir Osmangazi University (Other)
Responsible Party: Eskisehir Osmangazi University, Department of Chest Diseases, Intensive Care Unit, Eskisehir Osmangazi University
Other Study IDs: HAP-OU-isolation
Record Dates: First submitted 2010-11-30; First posted 2010-12-01 (Estimated); Last update posted 2010-12-01 (Estimated); Status verified 2004-01

CONDITIONS: Pneumonia; Intensive Care Unit
Keywords: pneumonia; ICU; isolation room; clinical epidemiology; infection control
MeSH Terms: conditions — Pneumonia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- hospital acquired pneumonia
- isolated rooms
  Interventions: Other: ward-type ICU
- ward-type ICU

INTERVENTIONS:
Other: ward-type ICU — frequency of hospital acquired pneumonia in the ICU
  Other Names: frequency of hospital acquired pneumonia in the ICU
  Groups: isolated rooms

SUMMARY:
This study will carry out in the ICU. Objectives of the study are to determine the frequency of HAP and the effect of isolated rooms on the frequency of pneumonia in the ICU.

DETAILED DESCRIPTION:
In the present study, it was aimed to determine the incidence, causative agents, antimicrobial resistance, and risk factors for lower respiratory tract infections in patients followed in the ICU for the last 4 years. The effect of reconfiguration from a ward-type ICU consisting one large room to an ICU with isolated rooms with two beds on the incidence of HAP was also determined.

ELIGIBILITY:
Inclusion Criteria:

* adult patients,
* admitted to the ICU

Exclusion Criteria:

* trauma, surgery or burned patients
* patients under 18

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All of the patients who had been admitted to the ICU during this period were included in the study
Sampling Method: Non-Probability Sample
Enrollment: 532 (Actual)
Dates: Start 2004-01; Primary Completion 2008-07 (Actual); Study Completion 2010-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Irfan Ucgun, As.Prof.Dr., Study Chair — Eskisehir Osmangazi University, Medical Faculty
Locations (3):
- Turkey (Türkiye) (3):
  - Eskisehir Osmangazi University, Eskişehir, Merkez
  - Osmangazi University, Eskişehir, Merkez
  - Eskisehir Osmangazi University, Eskişehir